CLINICAL TRIAL: NCT03469492
Title: Investigating the Role of the Polyol Pathway in the Central Nervous System Production of Fructose: an Intervention Study
Brief Title: Investigating the Role of the Polyol Pathway in the Central Nervous System Production of Fructose
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1602017151; 1K23DK109284-01 (NIH)
Record Dates: First submitted 2018-01-11; First posted 2018-03-19 (Actual); Results first posted 2023-02-02 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Hyperglycaemia (Diabetic)
MeSH Terms: conditions — Hyperglycemia | interventions — Insulin; Exercise; Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- type 2 diabetes mellitus (Active Comparator): Subjects with type 2 diabetes on insulin.
  Interventions: Drug: Insulin; Behavioral: exercise; Dietary Supplement: Dietary counseling
- type 1 diabetes mellitus (Active Comparator): Subjects with type 1 diabetes on insulin.
  Interventions: Drug: Insulin; Behavioral: exercise; Dietary Supplement: Dietary counseling

INTERVENTIONS:
Drug: Insulin — Insulin regimens will be adjusted on a weekly basis as needed to achieve a target blood glucose level.
Behavioral: exercise — Exercise in accordance to the guidelines established by the American Diabetes Association.
Dietary Supplement: Dietary counseling — Dietary counseling in accordance to the guidelines established by the American Diabetes Association.

SUMMARY:
To investigate whether longer-term improvement of glycemic control in poorly controlled diabetes patients with a 12-week intensified insulin treatment regimen will lead to decreased polyol pathway activity.

DETAILED DESCRIPTION:
Polyol pathway activity will decrease in diabetic individuals who undergo intensification of their insulin treatment regimens as reflected by lower baseline brain intracellular fructose levels and higher intracellular glutathione levels. Furthermore, following longer-term improved glycemic control, patients may also have down-regulation of the pathway as reflected by decreased production of intracellular fructose in response to hyperglycemic clamp.

ELIGIBILITY:
Inclusion Criteria:

* 15 Type 2 DM subjects with HbA1C > 7.5%
* 15 Type 1 DM subjects with HbA1C > 7.5%
* Age 18-60
* BMI ≥18 kg/m2
* Weight ≤ 285 pounds

Exclusion Criteria:

* Creatinine > 1.5 mg/dL, Hgb < 10 mg/dL, ALT > 2.5 X ULN,
* untreated thyroid disease,
* uncontrolled hypertension,
* known neurological disorders,
* untreated psychiatric disorders,
* malignancy,
* bleeding disorders,
* current or recent steroid use in last 3 months,
* illicit drug use;
* for women: pregnancy, actively seeking pregnancy, or breastfeeding; inability to enter
* MRI/MRS

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janice Hwang, MD, Principal Investigator — Section of Endocrinology
Locations (1):
- The Anylan Center, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Sanchez-Rangel E, Gunawan F, Jiang L, Savoye M, Dai F, Coppoli A, Rothman DL, Mason GF, Hwang JJ. Reversibility of brain glucose kinetics in type 2 diabetes mellitus. Diabetologia. 2022 May;65(5):895-905. doi: 10.1007/s00125-022-05664-y. Epub 2022 Mar 5. PMID 35247067

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Type 2 Diabetes Mellitus
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Type 2 Diabetes Mellitus
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.8 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 2
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 10 (8.2)
BMI [Mean (Standard Deviation); unit: kilograms/meter square] | 31.4 (6.1)
Weight [Mean (Standard Deviation); unit: kilograms] | 85 (21.2)
HbA1c [Mean (Standard Deviation); unit: mmol/mol] | 84.1 (16.2)
HbA1c [Mean (Standard Deviation); unit: percentage glycated hemoglobin] | 9.8 (1.4)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c Levels
Description: HbA1c levels measured by MRS scanning during a hyperglycaemic clamp. Result reported is the mean decrease in HbA1C. A decrease in HbA1c indicates improvement in brain glucose levels.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: mmol/mol
Arm/Group | Type 2 Diabetes Mellitus
Number analyzed (Participants) | 8
mmol/mol | 24.3 (15.3)
Statistical Analysis 1: Comparison: Type 2 Diabetes Mellitus; Test type: Superiority; p = 0.006, Regression, Linear

2. Secondary Outcome: Gluthathione
Description: baseline MRS scan to measure gluthathione
Time Frame: 0 weeks
Population: Data for this outcome not collected.
Arm/Group | Type 2 Diabetes Mellitus
Number analyzed (Participants) | 0

3. Secondary Outcome: Gluthathione
Description: MRS scan to measure gluthathione
Time Frame: 12 weeks
Population: Data for this outcome not collected.
Arm/Group | Type 2 Diabetes Mellitus
Number analyzed (Participants) | 0

4. Secondary Outcome: Plasma Glucose
Description: MRS scan to measure plasma glucose
Time Frame: 0 weeks
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Type 2 Diabetes Mellitus
Number analyzed (Participants) | 8
mmol/l | 1.07 (.23)

5. Secondary Outcome: Plasma Glucose
Description: MRS scan to measure plasma glucose
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Type 2 Diabetes Mellitus
Number analyzed (Participants) | 8
mmol/l | 0.88 (0.35)
Statistical Analysis 1: Comparison: Type 2 Diabetes Mellitus; Test type: Superiority; p = 0.266, Mixed Models Analysis

6. Secondary Outcome: Plasma Fructose
Description: MRS scan to measure plasma fructose
Time Frame: 0 weeks
Population: Data for this outcome not collected.
Arm/Group | Type 2 Diabetes Mellitus
Number analyzed (Participants) | 0

7. Secondary Outcome: Plasma Fructose
Description: MRS scan to measure plasma fructose
Time Frame: 12 weeks
Population: Data for this outcome not collected.
Arm/Group | Type 2 Diabetes Mellitus
Number analyzed (Participants) | 0

8. Secondary Outcome: Plasma Insulin
Description: MRS scan to measure plasma insulin
Time Frame: 0 weeks
Measure: Mean (Standard Deviation); unit: μU/ml
Arm/Group | Type 2 Diabetes Mellitus
Number analyzed (Participants) | 8
μU/ml | 31 (26)
Statistical Analysis 1: Comparison: Type 2 Diabetes Mellitus; Test type: Superiority; p = 0.20, Mixed Models Analysis

9. Secondary Outcome: Plasma Insulin
Description: MRS scan to measure plasma insulin
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: μU/ml
Arm/Group | Type 2 Diabetes Mellitus
Number analyzed (Participants) | 8
μU/ml | 38 (29)
Statistical Analysis 1: Comparison: Type 2 Diabetes Mellitus; Test type: Superiority; p = 0.25, Mixed Models Analysis

10. Other Pre Specified Outcome: Optional Hyperglycemic Clamp
Description: Hyperglycemic clamp administered to measure glucose levels. Data represented is the number of participants the clamp was used on successfully.
Time Frame: upon enrollment
Measure: Number; unit: participants
Arm/Group | Type 2 Diabetes Mellitus
Number analyzed (Participants) | 8
participants | 8

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the course of the study from baseline up to 24 months.
Arm/Group | Type 2 Diabetes Mellitus
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-14): https://cdn.clinicaltrials.gov/large-docs/92/NCT03469492/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-14): https://cdn.clinicaltrials.gov/large-docs/92/NCT03469492/ICF_001.pdf